CLINICAL TRIAL: NCT06687525
Title: Alcohol and the Social Brain: an Alcohol-Administration Hyperscanning Study
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Other Study IDs: 2R01AA025969 (NIH)
Record Dates: First submitted 2024-08-26; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder; Alcohol Intoxication; Alcohol; Harmful Use; Alcoholism; Binge Drinking
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcoholic Intoxication; Binge Drinking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, the investigators aim to capture inter- and intra-brain mechanisms underlying alcohol reward in novel social context.

DETAILED DESCRIPTION:
Objective: Alcohol's ability to boost mood in the face of stress is perhaps its most notoriously addictive property, long held by researchers to be of critical importance for understanding alcohol use disorder (AUD) etiology. Yet, while most real-world alcohol consumption occurs in social settings, in the context of laboratory studies, participants have almost always consumed alcohol alone. The discrepancy between real-world and laboratory contexts emerges as particularly stark in the neuroimaging literature, where no alcohol-administration study to date has incorporated in-vivo social context. In this first alcohol-administration study to leverage EEG hyperscanning methods, the investigators aim to capture inter- and intra-brain mechanisms underlying alcohol reward in novel social context.

Specifically, this study aims to characterize the mechanisms driving social reward from alcohol in the context of stress and elucidate the role of social processes and novel social context in driving problem drinking.

Study Population: Participants will consist of 240 regular drinkers, aged 21-30, with no reported history of severe alcohol use disorder.

Design: In the laboratory arm of the study, individuals will be randomly assigned to consume either a moderate dose of alcohol or a control beverage in stranger dyads. Participants will engage in both structured and unstructured tasks aimed at assessing social engagement and threat sensitivity. EEG and ERP data will be collected from both participants simultaneously. In the ambulatory study arm, participants will wear transdermal sensors to assess BAC and will further provide information about their mood and their social contexts in response to random prompts.

Outcome Measures: Primary outcome measures include EEG measures of inter-brain entrainment as well as ERP metrics derived from task contexts (both players and observers). Additional outcomes include measures of positive mood, negative mood, and social bonding. Finally, drinking behaviors will be assessed via transdermal ambulatory alcohol sensors and longitudinal self-reports of drinking.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 and 30
* Regularly consumes alcohol

Exclusion Criteria:

* History of adverse reaction to the amount of beverage employed in the study
* Have a history of major problems associated with alcohol
* Take medications that could adversely interact with alcohol
* Have medical conditions that contraindicate alcohol administration
* Individuals with a history of skull fractures or who indicate discomfort with EEG procedures used
* Female participant is pregnant or trying to become pregnant

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy regular drinkers aged 21-30
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Inter-brain entrainment | During active laboratory beverage manipulation exposure (during or immediately after beverage administration, at which time participants in the alcohol condition will register a positive BAC)
  The association between dyad-members EEG signals during the hyperscanning task
Feedback-related negativity | During active laboratory beverage manipulation exposure (during or immediately after beverage administration, at which time participants in the alcohol condition will register a positive BAC)
  An ERP component calculated from a time-estimation task
Ambulatory Drinking | 14 days
  Drinking behavior assessed outside the laboratory using ambulatory assessment
Longitudinal Drinking Problems | Up to 24 months post-baseline
  Drinking assessed at longitudinal follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Catharine E Fairbairn, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is being shared on the National Institute of Mental Health Data Archive
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Sayette MA, Creswell KG, Dimoff JD, Fairbairn CE, Cohn JF, Heckman BW, Kirchner TR, Levine JM, Moreland RL. Alcohol and group formation: a multimodal investigation of the effects of alcohol on emotion and social bonding. Psychol Sci. 2012 Aug 1;23(8):869-78. doi: 10.1177/0956797611435134. Epub 2012 Jul 3. PMID 22760882
- [Background] Fairbairn CE, Sayette MA. A social-attributional analysis of alcohol response. Psychol Bull. 2014 Sep;140(5):1361-82. doi: 10.1037/a0037563. PMID 25180806
- [Background] Fairbairn CE, Kang D, Federmeier KD. Alcohol and Neural Dynamics: A Meta-analysis of Acute Alcohol Effects on Event-Related Brain Potentials. Biol Psychiatry. 2021 May 15;89(10):990-1000. doi: 10.1016/j.biopsych.2020.11.024. Epub 2020 Dec 11. PMID 33579536